CLINICAL TRIAL: NCT02305836
Title: The Effect of Electroacupuncture Combined With Donepezil on Cognitive Function in Alzheimer's Disease Patients: Study Protocol for a Randomized Controlled Trial
Brief Title: Effect of Electroacupuncture Combined With Donepezil for Treating Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Weina Peng, Dean of Acupuncture Department of Guangan'men Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2014S291
Record Dates: First submitted 2014-11-13; First posted 2014-12-03 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Cognitive Impairment
Keywords: Electroacupuncture; Donepezil; Alzheimer's disease; Randomized controlled trial
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Acupuncture Therapy; Electroacupuncture; Donepezil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture combined with donepezil (Experimental): Every session will last for 30 minuets and will be given every other day. There are 36 sessions for each participant in all (3 session per week, 12 weeks).
  Interventions: Procedure: acupuncture
- donepezil (Active Comparator): Donepezil will be given once daily before bed-time for the first 4-6 weeks. Based on the treatment effect, the dosage may be increased to 10 mg once daily before bed-time for the next 6-8 weeks. Donepezil will be taken for continuous 24 weeks. The full course of treatment is 36 weeks.
  Interventions: Drug: donepezil

INTERVENTIONS:
Procedure: acupuncture — For GV16, the needle in length of 25mm will be inserted obliquely and downward towards mandibular direction slowly to a depth of 0.5. And the needle will be pulled out after "de qi" without being retained. For Shang Yintang, GV20 and GV24, the needle will be inserted with a 30°angle to a depth of about 0.5 cun to the subperiosteum until the patients have a strong sense that the needle is being heavily pressed. For EX-HN5 and KI 4 in both sides, the needle will be outward and obliquely inserted to the same depth of 1 cun and the needle will be manipulated with an even lifting and thrusting method to make the patients feel soreness and distention. The electric stimulator will be put on GV20, GV24 and EX-HN5 in both sides with a spare-dense wave, 10/50 Hz, 0.5-5.0 mA. The current intensity will be increased until the patients can not stand.
  Other Names: electroacupuncture
  Arms: Electroacupuncture combined with donepezil
Drug: donepezil — cholinesterase inhibitors (ChE-Is)
  Other Names: Aricept
  Arms: donepezil

SUMMARY:
A prospective randomized controlled trial aimed at assessing if electroacupuncture (EA) combined with donepezil is more effective than donepezil for improving the cognitive function of AD patients. The hypothesis of this study is as follow:

* Is the short-term effect of EA combined with donepezil better than donepezil on improving cognitive function of patients with Alzheimer's disease after 12 weeks' treatment?
* Whether the effect of EA combined with donepezil on improving cognitive function can last until the end of 6 months' follow-up?

DETAILED DESCRIPTION:
* Patient registry: Participants experiencing cognitive impairment will be recruited will be recruited at Guang'anmen Hospital, Beijing, China, via web or posters. A neurologist will make the diagnosis. Randomization will be performed by the pharmacological assessment center at Guang'anmen Hospital.
* Sample size: The calculation of sample size is based on the primary outcome that the change from baseline in ADAS-cog. According to previous studies [26], 39% of patients showed an improvement of at least 4 points on the ADAS-cog after treating by donepezil. We estimated the rate 39% in the donepezil group and 55% in the EA combined with donepezil group. 304 participants were needed to provide 80% power at a significant level of 5% using analysis of variance. The total sample size required for the study is 334 (167 each group) assuming a 10% loss to follow-up.
* Quality control

  1. Investigators participating in this trial will take a strict course about the process of randomization, manipulation of electroacupuncture, selection of patients, the whole process of this trial and request for filling out case report form in order to improve the internal consistency of observation between different researchers.
  2. The process of randomization will be under a rigorous control.
  3. This trial has a specific inclusion and exclusion criteria.
  4. Both outcome assessors and statisticians will be blinding.
  5. Patients will sign the informed consent voluntarily and a good relationship between researchers and patients will be established in order to improve patients' compliance. Participants will have a detailed record of the contact information easy for follow-up.
  6. The standard of the drugs, acupuncture apparatus, inspection equipment are consistent for the patients in the two groups.
* Outcome assessment, completion of case report forms and data management will be under a rigorous supervision.

ELIGIBILITY:
Inclusion Criteria:

Participants meeting all of the following criteria will be included in this trial: 1) the diagnostic criteria of Neurological Communicative Disorders and Stroke and the Alzheimer Disease and Related Disorders Association (NINCDS-ADRDA) or the Operational Criteria for the Diagnosis of Alzheimer's disease (OCDAD), 2) aged between 60-85 years, 3) cognitive impairment based on the scores of the Chinese version of the Mini Mental State Examination (MMSE) (illiteracy group ≤19, primary school group ≤22, junior high school and high school group ≤23, and well-educated group ≤26), 4) absence of depression (via an emotional assessment), 5) Magnetic Resonance Imaging (MRI) confirmation of atrophy of the hippocampus or the medial temporal lobe volume, 6) the Medial Temporal Lobe Atrophy Rating Scale (MTA-scale) score (≥ 2 for those under 75 years, and ≥ 3 for those over 75 years).

Exclusion criteria:

Participants meeting any one of the following criteria will be excluded from this trial: 1) Cognitive impairment caused by other factors (e.g. vascular dementia, dementia with Lewy's bodies, frontotemporal dementia, hormone or metabolic abnormalities, hypothyroidism, folic acid or vitamin B12 deficiency, delirium or other mental and emotional disorders [such as schizophrenia and depression]), 2) a serious heart condition, hepatic disease, renal system disease, hematopoietic system disease, or malnutrition of the whole body, 3) aphasia or decreased vision that is severe, blindness, disturbance of consciousness, or participants who cannot cooperate with the related examinations due to physical disability, 4) anticoagulant treatments such as warfarin or heparin, 5) use of pacemakers or participants too afraid of acupuncture, or 6) acupuncture or donepezil treatment in the past 30 days.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
change of total ADAS-cog score from baseline | week 12 ± 3 days
  The maximum score of ADAS-cog is 70 including 15 items of cognitive dysfunction assessment. The higher values indicate higher degree of deficit.

SECONDARY OUTCOMES:
change of total MMSE score from baseline | week 12 ± 3 days
  MMSE score are commonly used for estimating the severity of cognitive impairment with maximum score of 30. The questions in this scale included orientation to time, orientation to place, attention and calculation, recall of three words and visual construction.
change of total MMSE score from baseline | week 36 ± 3 days
change of total ADCS-ADL score score from baseline | week 12 ± 3 days
  ADCS-ADL score contains 19 domains about assessment of basic and operational ability of daily living.
change of total ADCS-ADL score score from baseline | week 36 ± 3 days
change of total QoL-AD score score from baseline | week 12 ± 3 days
  QOL-AD score which includes physical health, mental health, social and financial assessment and QOL domains is completed by both patients and caregivers.
change of total QoL-AD score score from baseline | week 36 ± 3 days
change of total ADAS-cog score from baseline | week 36 ± 3 days

OTHER OUTCOMES:
Safety related evaluation of electroacupuncture as measured by number of participants with adverse events. | from week 1 up to week 12
  Adverse reactions related with electroacupuncture such as fainting, haematomas, and local infection, the score of VAS more than 8 and other symptoms lasting for 1 hour or longer after acupuncture will be recorded in a designed table.
Safety related evaluation of Donepezil as measured by number of participants with adverse events. | from week 1 up to week 36
  Adverse reactions such as fasciculation, diarrhoea, fatigue, nausea, vomit and insomnia related to Donepezil will be be recorded in a designed table.

CONTACTS AND LOCATIONS:
Overall Officials: Weina Peng, Study Director — Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences
Locations (1):
- Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Peng W, Zhou J, Xu M, Feng Q, Bin L, Liu Z. The effect of electroacupuncture combined with donepezil on cognitive function in Alzheimer's disease patients: study protocol for a randomized controlled trial. Trials. 2017 Jul 3;18(1):301. doi: 10.1186/s13063-017-2052-y. PMID 28673322